CLINICAL TRIAL: NCT01241058
Title: Belgian Registry of Pediatric Crohn's Disease
Brief Title: Registry of Pediatric Patients Diagnosed With Crohn's Disease in Belgium
Acronym: Belcro
Status: Completed | Type: Observational
Sponsor: Gigi Veereman (Other)
Responsible Party: Sponsor-Investigator, Gigi Veereman, MD PHD Pediatric Gastroenterologist, Belgian Society for Pediatric Gastroentrology Hepatology and Nutrition
Organization: Belgian Society for Pediatric Gastroentrology Hepatology and Nutrition (Other)
Other Study IDs: Bespghan
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Description of Disease Course, Disease Fenotype, Medication, Safety, Analysis for Possible Associations
Keywords: pediatrics, crohn's disease, disease course, therapy
MeSH Terms: conditions — Crohn Disease; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A registry of pediatric patients (under 18 yrs of age) diagnosed with Crohn's disease was created in Belgium. Over a 2 year period 257 patients are included. These patients will be follow up prospectively during 5 years. Demographic data, family history, disease presentation and disease course including medication are registered in CRF's.

ELIGIBILITY:
Inclusion Criteria:

1-18 yrs old belgian Crohn s disease informed consent

Exclusion Criteria:

no informed consent

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: subjects under 18 yrs of age diagnosed with Crohn's disease, living in Belgium
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2008-05; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
disease course | 5 years
  describe patient characteristics, disease fenotype and course

CONTACTS AND LOCATIONS:
Locations (1):
- Bespghan, Leuven, Brabant, Belgium

REFERENCES:
- [Result] Van Biervliet S, Smets F, Hofmann I, Degreef E, Hauser B, Bontems P, Vande Velde S, Arts W, Paquot I, Alliet P, Bossuyt P, Louis E, Baert F, Bauraind O, Rahier JF, Veereman G. The course of anaemia in children and adolescents with Crohn's disease included in a prospective registry. Int J Colorectal Dis. 2015 Jan;30(1):51-6. doi: 10.1007/s00384-014-2042-4. Epub 2014 Oct 30. PMID 25354967
- [Result] De Greef E, Maus B, Smets F, Van Biervliet S, John JM, Van Steen K, Veereman G; IBD working group of the Belgian Society of Pediatric Gastroenterology, Hepatology and Nutrition (BeSPGHAN); Belgian IBD Research and Development (BIRD). Diagnosing and treating pediatric Crohn's disease patients: is there a difference between adult and pediatric gastroenterologist's practices ? Results of the BELCRO cohort. Acta Gastroenterol Belg. 2014 Mar;77(1):25-9. No abstract available. PMID 24761688
- [Result] De Greef E, Mahachie John JM, Hoffman I, Smets F, Van Biervliet S, Scaillon M, Hauser B, Paquot I, Alliet P, Arts W, Dewit O, Peeters H, Baert F, D'Haens G, Rahier JF, Etienne I, Bauraind O, Van Gossum A, Vermeire S, Fontaine F, Muls V, Louis E, Van de Mierop F, Coche JC, Van Steen K, Veereman G; IBD working group of the Belgian Society of Pediatric Gastroenterology, Hepatology and Nutrition (BeSPGHAN); Belgian IBD Research and Development. Profile of pediatric Crohn's disease in Belgium. J Crohns Colitis. 2013 Dec;7(11):e588-98. doi: 10.1016/j.crohns.2013.04.016. Epub 2013 May 9. PMID 23664896
- [Result] Alliet P, Desimpelaere J, Hauser B, Janssens E, Khamis J, Lewin M, De Greef E, Smets F, Paquot I, Veereman G, Souverijns G; Belgian IBD working group of BeSPGHAN. MR enterography in children with Crohn disease: results from the Belgian pediatric Crohn registry (Belcro). Acta Gastroenterol Belg. 2013 Mar;76(1):45-8. PMID 23650782
- [Derived] De Greef E, Hoffman I, Smets F, Van Biervliet S, Bontems P, Hauser B, Paquot I, Alliet P, Arts W, Dewit O, De Vos M, Baert F, Bossuyt P, Rahier JF, Franchimont D, Vermeire S, Fontaine F, Louis E, Coche JC, Veereman G; IBD working group of BESPGHAN, BIRD. Paediatric Crohn Disease: Disease Activity and Growth in the BELCRO Cohort After 3 Years Follow-up. J Pediatr Gastroenterol Nutr. 2016 Aug;63(2):253-8. doi: 10.1097/MPG.0000000000001132. PMID 26835906